CLINICAL TRIAL: NCT06003465
Title: A Relative Bioavailability Study to Compare the Pharmacokinetics of LY3437943 Administered Subcutaneously by a Test Device (Test Formulation) Versus Reference Device (Reference Formulation) in Healthy Participants
Brief Title: A Research Study Looking at Similarity Between LY3437943 Versions for Different Injection Devices
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18530; J1I-MC-GZBX (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-08-16; First posted 2023-08-22 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — retatrutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- LY3437943 - Test (Experimental): A single dose of LY3437943 administered by subcutaneous (SC) injection via a test device (test formulation)
  Interventions: Drug: LY3437943; Device: Test
- LY3437943 - Reference (Active Comparator): A single dose of LY3437943 administered by SC injection via a reference device (reference formulation)
  Interventions: Drug: LY3437943; Device: Reference

INTERVENTIONS:
Drug: LY3437943 — Administered SC
Device: Test — Used to administer LY3437943 SC
  Arms: LY3437943 - Test
Device: Reference — Used to administer LY3437943 SC
  Arms: LY3437943 - Reference

SUMMARY:
The main purpose of this study is to look at the amount of the study drug, LY3437943, that gets into the blood stream and how long it takes the body to get rid of it when given using two different devices. The study will also evaluate the safety and tolerability of LY3437943 and information about any side effects experienced will be collected. For each participant, the total duration of the study will be approximately 16 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant females as determined by medical history, physical examination, and other screening procedures
* Body mass index (BMI) between 18.5 and 32.0 kilograms per meter squared (kg/m²), inclusive
* Have clinical laboratory test results, blood pressure and pulse rate that are acceptable for the study
* Are agreeable to receiving study treatment by injections under the skin
* Males who agree to use highly effective/effective methods of contraception and women not of childbearing potential (postmenopausal or oophorectomized)

Exclusion Criteria:

* Have or used to have health problems that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Smoke more than the equivalent of 10 cigarettes per day
* Is a known user of drugs of abuse
* Have known allergies to LY3437943 or related compounds

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3437943 | Predose up to 43 days postdose
  PK: Cmax of LY3437943
PK: Area Under the Plasma Concentration Versus Time Curve from Zero to T, Last Time Point (AUC[0-tlast]) of LY3437943 | Predose up to 43 days postdose
  PK: AUC[0-tlast] of LY3437943
PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3437943 | Predose up to 43 days postdose
  PK: AUC(0-∞) of LY3437943

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - Qps-Mra, Llc, Miami, Florida
  - ICON Early Phase Services, San Antonio, Texas
  - ICON, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No